CLINICAL TRIAL: NCT01055171
Title: Treatment Implications of Trauma Memory Modulation for PTSD & Alcohol Dependence
Brief Title: Neuromodulation of Trauma Memories in PTSD & Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19489; 1RC1AA019019-01 (NIH)
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2012-09

CONDITIONS: Alcohol Dependence; PTSD
Keywords: alcohol dependence; PTSD; propanolol; craving; beta-block; cue exposure; addiction; memory; trauma; addictive behavior
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Behavior, Addictive; Wounds and Injuries | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Active Comparator): Patients will receive Propranolol in this condition.
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Patient to receive placebo in this condition.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 40 mg; Single Administration.
  Arms: Propranolol
Drug: Placebo — 40 mg; Single Dose.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of propranolol versus placebo on craving, distress and cue reactivity to trauma and alcohol cues.

DETAILED DESCRIPTION:
Summary and Synthesis: Epidemiological studies have established the occurrence of high rates of AD in persons with PTSD. Likewise, studies of alcohol/drug abuse treatment seekers have documented high rates of trauma exposure and PTSD. The high prevalence of PTSD/AD comorbidity is the cause of enormous human suffering, most of which either goes untreated or is resistant to treatment efforts. Both theory and research concerning the interface between these two disorders suggests that PTSD is associated with the initiation of excessive alcohol use and/or the development of AD by way of an escape/avoidance behavioral mechanism wherein escalating alcohol use is reinforced by its ability to dampen the negative emotions and arousal associated with PTSD. If PTSD is often a primary cause of the initiation and maintenance of AD, then clinical interventions that primarily impact PTSD should lead to significant improvements in craving for, and use of, alcohol. The findings of two recent treatment studies offer especially compelling support for this expectation. Drawing on both basic neuroscience research and a developing body of suggestive clinical/applied research, we were led to consider if the putative memory modulating properties of the adrenergic antagonist propranolol might have therapeutic benefits for PTSD/AD comorbid individuals. Thus, the proposed study will test the hypothesis that the strategic administration of propranolol coupled with the elicitation/retrieval of trauma-related memories will dampen emotional distress, alcohol craving and cue reactivity during subsequent exposure to trauma- and alcohol-related cues. A two-week follow-up laboratory session and clinical assessment will permit us to evaluate whether treatment benefits are maintained over time and if there are any changes in alcohol use and PTSD symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet DSM-IV criteria for current alcohol dependence
* Participants must have experienced criminal victimization
* Use of birth control by female participants
* Live within a 50-mile radius of research site
* Consent to remain abstinent of all drugs and alcohol for 24 hours prior to patient admission and follow-up
* Consent to random assignment to propanol or placebo
* Individuals must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.

Exclusion Criteria:

* Women who are pregnant, nursing or are of childbearing potential and not using birth control.
* Evidence or history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal or neurological disease
* Significant liver impairment
* Currently taking anti-arrhythmic agents, psychostimulants or other agents known to interfere with heart rate and skin conductance monitoring.
* Known or suspected hypersensitivity to propanol
* Individuals taking medication that could adversely interact with the study medication, including the following: albuterol, insulin or significant inhibitors of CYP2D6
* Individuals with bronchial asthma or chronic obstructive pulmonary disease
* Prospective participants will be excluded if they are currently receiving exposure-based therapy for PTSD.
* Individuals with a history of or current psychotic disorder.
* Individuals with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect cortisol levels.
* Individuals receiving synthetic glucocorticoid therapy, any exogenous therapy, or treatment with other agents that interfere with HPA axis function within one month of the time of testing.
* Individuals with resting heart rates less than 55 bpm.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Saladin, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered enrolled if they completed both the retrieval and testing procedure (44).
Groups:
- Propranolol: Patients will receive Propranolol in this condition.
  Propranolol : 40 mg; Single Administration.
  The subjects analyzed who received propranolol were those that received the medication and completed both the test and retrieval sessions (Test Day 1 and 2).
- Placebo: Patient to receive placebo in this condition.
  Placebo : 40 mg; Single Dose.
  The subjects analyzed who received placebo were those that received the sugar pill and completed both the test and retrieval sessions (Test Day 1 and 2)
Period: Overall Study
Arm/Group | Propranolol | Placebo
Started | 29 (Randomized to receive medication.) | 28 (Randomized to receive placebo.)
Retrieval Completion | 25 (Received the medication and completed the retrieval session.) | 24 (Received the sugar pill and completed the retrieval session.)
Test Procedure Completion | 21 (Received the medication and completed the first test session.) | 23 (Received the placebo and completed the first test session.)
Completed | 18 (Received the medication and completed all visits including the one-week follow-up.) | 21 (Received the sugar pill and completed all visits including the one-week follow-up.)
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Population: Urn randomization was used to assign participants to the propranolol vs. placebo condition while balancing treatment assignment on gender and age (less than 35 or equal to or greater than 35 years of age).
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Customized [Number; unit: Participants]
  Greater than or equal to 35 years | 14 | 17 | 31
  Less than 35 years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Retrieval Session Distress Scores (Session 1)
Description: Found by using our Single Item Distress (SID) scale. A study team member asks the participant to verbally report the level of distress they were experiencing using values between 0 and 100, with 0 representing no distress and 100 extreme distress.
Time Frame: Multiple times throughout cue exposure during retrieval session (Session 1)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 21 | 23
units on a scale | 54.5 (26.8) | 73.9 (20.9)

2. Primary Outcome: Retrieval Session Craving Scores (Session 1)
Description: Found by using our Single Item Craving (SIC) scale. A study team member asks the participant to verbally report the level of craving they were experiencing using values between 0 and 100, with 0 representing no craving and 100 extreme craving for alcohol.
Time Frame: Multiple times throughout cue exposure during retrieval session (Session 1)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 21 | 23
units on a scale | 49.1 (31.3) | 71.6 (20.4)

3. Primary Outcome: Test Session Distress Scores (Session 2)
Description: as for outcome 1
Time Frame: Multiple times throughout cue exposure during test session (Session 2)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 21 | 23
units on a scale | 35.1 (3.7) | 48.0 (3.5)

4. Primary Outcome: Test Session Craving Scores (Session 2)
Description: as for outcome 2
Time Frame: Multiple times throughout cue exposure during test session (Session 2)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 21 | 23
units on a scale | 51.0 (3.7) | 53.9 (3.5)

5. Secondary Outcome: Proportion of Drinking Days
Description: Proportion of drinking days from 90 days prior to the screening to the follow-up period.
Time Frame: 90 days prior to participation in study up to 2-week follow up session (Session 3)
Measure: Mean (Standard Error); unit: Drinking days
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 21 | 23
Drinking days | 42.2 (6.4) | 45.9 (6.8)

ADVERSE EVENTS:
Arm/Group | Propranolol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

LIMITATIONS AND CAVEATS:
Lack of a "no retrieval" control group. Lack of determination of plasma propranolol levels following the medicated retrieval session. The sample size was insufficient to assess the more distal effects at 1-week follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No